CLINICAL TRIAL: NCT03434223
Title: Prospective Follow-up of Elderly Patients Undergoing Instrumented Lumbar Arthrodesis Supplemented by the Implanet Jazz System(TM)
Status: Terminated | Type: Observational
Why Stopped: Research has been discontinued - there will be no further data collection or analysis
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, H Francis Farhadi, MD, PhD, Assistant Professor, Ohio State University
Other Study IDs: 2016H0350
Record Dates: First submitted 2018-02-09; First posted 2018-02-15 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Spondylolisthesis; Spinal Stenosis; Degenerative Disease
MeSH Terms: conditions — Spondylolisthesis; Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Cohort

SUMMARY:
Establish a data repository of patients who have undergone single, two-, or three-level lumbar instrumented arthrodesis procedures supplemented by the Implanet Jazz System.

DETAILED DESCRIPTION:
To collect and organize data into a repository from the Principal Investigator's and other Site Investigators' elderly patients (aged ≥ 60 years) who are undergoing single, two-level, or three-level lumbar instrumented arthrodesis procedures supplemented by the Implanet Jazz SystemTM at participating centers. This device is designed to provide a stable interface between spinal constructs and the rods; it can be secured around vertebral structures (such as the lamina, transverse or spinous processes) from T1 to L5 and is intended to provide temporary stabilization as a bone anchor during the development of a solid body fusion. Of note, these patients will receive the supplemental support of the Implanet Jazz Sublaminar Band as their clinical standard of care deems necessary and separately from study participation.

Clinical data will be collected as indicated at 6 weeks, as well as 3, 6, 12, 24, 36, 48, and 60 months post-operatively in the database.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are candidates for single, two- or three-level spinal arthrodesis surgery supplemented by the Implanet Jazz System
* Patients at least 60 years of age.

Exclusion Criteria:

* Patients under the age of 60 years old are excluded.

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are candidates for single, two- or three-level spinal arthrodesis surgery supplemented by the Implanet Jazz System
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2016-12-29 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
Number of patients who have undergone lumbar instrumented arthrodesis procedures supplemented by the Implanet Jazz System | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: H. Francis Farhadi, MD, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No